CLINICAL TRIAL: NCT01968057
Title: A Study to Investigate the Effect of Ciclosporin on the Pharmacokinetics of Baricitinib (LY3009104) in Healthy Subjects
Brief Title: A Study of Baricitinib and Ciclosporin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14605; I4V-MC-JAGH (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — baricitinib; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baricitinib (Experimental): Single oral dose of 4 milligrams (mg) baricitinib on Day 1
  Interventions: Drug: Baricitinib
- Baricitinib + Ciclosporin (Experimental): Single oral dose of 4 mg baricitinib co-administered with a single oral dose of 600 mg ciclosporin on Day 4
  Interventions: Drug: Baricitinib; Drug: Ciclosporin

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
Drug: Ciclosporin — Administered orally
  Arms: Baricitinib + Ciclosporin

SUMMARY:
The purpose of this study is to determine the effects of ciclosporin on the amount of baricitinib that is absorbed into the blood stream and the time it takes to remove baricitinib from the body. The study will also look at how well-tolerated and safe baricitinib is, when given alone and in combination with ciclosporin. Side effects will be documented. The study will last approximately 6 days from the first dose to the end of the study (not including screening or follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Male participants: agree to use 2 reliable methods of birth control with female partners of childbearing potential during the study and for at least 3 months following the last dose of study drug
* Female participants: women not of childbearing potential due to surgical sterilization confirmed by medical history, or menopause
* Have a body mass index of 18.0 to 29.0 kilograms per meter squared (kg/m^2), inclusive
* Have clinical laboratory test results within the normal reference range
* Have normal renal function
* Have normal blood pressure and pulse rate

Exclusion Criteria:

* Are currently enrolled in a clinical trial involving a study drug or off-label use of a drug or device, or are concurrently enrolled in any other type of medical research
* Have completed or discontinued within the last 90 days from a clinical trial involving a study drug
* Are participants who have previously completed or withdrawn from this study or any other study investigating baricitinib, and have previously received baricitinib
* Have known allergies to baricitinib, ciclosporin, related compounds, or any components of the baricitinib or ciclosporin formulations, or history of significant atopy
* Have an abnormality in the 12-lead electrocardiogram (ECG)
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Have a current or recent history of a clinically significant bacterial, fungal, parasitic, viral (not including rhinopharyngitis), or mycobacterial infection
* Have had symptomatic herpes zoster or herpes simplex infection within 90 days prior to the first dose
* Have an absolute neutrophil count (ANC) less than 2 × 10^9 cells/liter(L) [2000 cells/microliter (μL)] at screening or day prior to first dose of study drug
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C infection and/or positive hepatitis C antibody
* Show evidence of hepatitis B infection and/or positive hepatitis B surface antigen
* Have a history of active tuberculosis within the last 5 years
* Are women who are lactating or pregnant
* Have been exposed to a live vaccine within 12 weeks prior to the first dose or expected to need/receive a live vaccine (including herpes zoster vaccination) during the course of the study
* Intend to use over-the-counter or prescription medication (including salicylate drugs) and/or herbal supplements within 14 days prior to dosing and during the study or intended use of vitamin supplements from Day 1 until discharge from the Clinical Research Unit (CRU)
* Have consumed or intend to consume grapefruit, Seville oranges, or products containing these fruits within 7 days prior to the first dose and until discharge from the CRU
* Have donated or lost blood of more than 500 milliliters (mL) within the last 3 months
* Have an average weekly alcohol intake that exceeds 28 units per week (males) and 21 units per week (females), or are unwilling to stop alcohol consumption from 48 hours prior to the first dose until discharge from the CRU at the end of Period 2
* History of, in the opinion of the investigator, excessive methylxanthine use within the previous 6 months, such as greater than (>) 6 cups of coffee (or equivalent) per day
* Currently smoke more than 10 cigarettes per day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, 2-period, fixed-sequence study.
Groups:
- Baricitinib + Ciclosporin: 4 milligrams (mg) baricitinib administered orally on Day 1 of Period 1.
  4 mg baricitinib co-administered with 600 mg ciclosporin on Day 4 of Period 2.
Period: Period 1 (Day 1 to Predosing Day 4)
Arm/Group | Baricitinib + Ciclosporin
Started | 18
Received Baricitinib | 18
Completed | 18
Not Completed | 0
Period: Period 2 (At Dosing Day 4 to Day 7)
Arm/Group | Baricitinib + Ciclosporin
Started | 18
Received Baricitinib + Ciclosporin | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Baricitinib + Ciclosporin: 4 mg baricitinib administered orally on Day 1 of Period 1.
  4 mg baricitinib co-administered with 600 mg ciclosporin on Day 4 of Period 2.
Arm/Group | Baricitinib + Ciclosporin
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 18

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Baricitinib
Time Frame: Days 1 and 4: predose of baricitinib, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 and 72 hours postdose
Population: All enrolled participants who received study drug (baricitinib in Period 1 and baricitinib + ciclosporin in Period 2) and had PK data to calculate Cmax of baricitinib.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- Baricitinib: 4 mg baricitinib administered orally on Day 1 of Period 1.
- Baricitinib + Ciclosporin: 4 mg baricitinib co-administered with 600 mg ciclosporin on Day 4 of Period 2.
Arm/Group | Baricitinib | Baricitinib + Ciclosporin
Number analyzed (Participants) | 18 | 18
nanograms/milliliter (ng/mL) | 36.2 (25) | 35.8 (22)

2. Primary Outcome: PK: Area Under the Concentration Curve From Time Zero to Infinity [AUC (0-∞)] of Baricitinib
Time Frame: Days 1 and 4: predose of baricitinib, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 and 72 hours postdose
Population: All enrolled participants who received study drug (baricitinib in Period 1 and baricitinib + ciclosporin in Period 2) and had PK data to calculate AUC (0-∞) of baricitinib.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | Baricitinib | Baricitinib + Ciclosporin
Number analyzed (Participants) | 18 | 18
nanograms*hour/milliliter (ng*h/mL) | 241 (24) | 311 (26)

3. Primary Outcome: PK: Time of Maximum Observed Drug Concentration (Tmax) of Baricitinib
Time Frame: Days 1 and 4: predose of baricitinib, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 and 72 hours postdose
Population: All enrolled participants who received study drug (baricitinib in Period 1 and baricitinib + ciclosporin in Period 2) and had PK data to calculate Tmax of baricitinib.
Measure: Median (Full Range); unit: hours
Arm/Group | Baricitinib | Baricitinib + Ciclosporin
Number analyzed (Participants) | 18 | 18
hours | 1.00 [0.50 to 1.00] | 2.00 [0.50 to 4.00]

ADVERSE EVENTS:
Time Frame: Baseline through study completion (up to Day 14).
Groups:
- Baricitinib: 4 mg baricitinib administered orally on Day 1 of Period 1.
  Adverse events are reported from baseline through predose on Day 4.
- Baricitinib + Ciclosporin: 4 mg baricitinib co-administered with 600 mg ciclosporin on Day 4 of Period 2.
  Adverse events are reported from postdose on Day 4 up to Day 14.
Arm/Group | Baricitinib | Baricitinib + Ciclosporin
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 9/18 | 15/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Baricitinib (N=18) | Baricitinib + Ciclosporin (N=18)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 8 (8)
Asthenia (General disorders) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2)
Feeling hot (General disorders) | 0 (0) | 6 (6)
Lethargy (General disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 2 (2)
Vessel puncture site anaesthesia (General disorders) | 0 (0) | 1 (1)
Vessel puncture site swelling (General disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 5 (5)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 8 (9)
Paraesthesia (Nervous system disorders) | 0 (0) | 3 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/3 (1) | 1/3 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin warm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days